CLINICAL TRIAL: NCT04268394
Title: A Phase 1, Open-label Study in Healthy Adult Subjects to Evaluate Effects of Cytochrome P450 Inhibition and Induction on the Pharmacokinetics of CC-99677 and the Effects of CC-99677 on the Pharmacokinetics of Digoxin, Metformin, Methotrexate, Midazolam, Rosuvastatin, and Sulfasalazine
Brief Title: A Study to Evaluate Potential Cytochrome P450 and Transporter Protein Interactions With CC-99677
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-99677-CP-002; U1111-1247-0554 (Registry Identifier: WHO); 2019-003523-38 (EudraCT Number)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Pharmacokinetics; Safety Tolerability; CC-99677
MeSH Terms: interventions — Methotrexate; Sulfasalazine; Itraconazole; Rifampin; Midazolam; Digoxin; Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: CC-99677 with Methotrexate and Sulfasalazine (Experimental): Fixed-sequence involving CC-99677 + Methotrexate 7.5 mg and sulfasalazine 1000 mg
  Interventions: Drug: CC-99677; Drug: Methotrexate; Drug: Sulfasalazine
- Part 2: CC-99677 with Itraconazole and Rifampin (Experimental): Fixed-sequence involving CC-99677 + Rifampin 600 mg and Itraconazole 200 mg
  Interventions: Drug: CC-99677; Drug: Itraconazole; Drug: Rifampin
- Part 3: CC-99677, Midazolam, Digoxin, Metformin, Rosuvastatin (Experimental): Fixed-sequence involving CC-99677 + Midazolam 2 mg, Digoxin 0.25 mg, Metformin 500 mg, and Rosuvastatin 10 mg.
  Interventions: Drug: CC-99677; Drug: Midazolam; Drug: Digoxin; Drug: Metformin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: CC-99677 — CC-99677
Drug: Methotrexate — Methotrexate
  Arms: Part 1: CC-99677 with Methotrexate and Sulfasalazine
Drug: Sulfasalazine — Sulfasalazine
  Arms: Part 1: CC-99677 with Methotrexate and Sulfasalazine
Drug: Itraconazole — Itraconazole
  Arms: Part 2: CC-99677 with Itraconazole and Rifampin
Drug: Rifampin — Rifampin
  Arms: Part 2: CC-99677 with Itraconazole and Rifampin
Drug: Midazolam — Midazolam
  Arms: Part 3: CC-99677, Midazolam, Digoxin, Metformin, Rosuvastatin
Drug: Digoxin — Digoxin
  Arms: Part 3: CC-99677, Midazolam, Digoxin, Metformin, Rosuvastatin
Drug: Metformin — Metformin
  Arms: Part 3: CC-99677, Midazolam, Digoxin, Metformin, Rosuvastatin
Drug: Rosuvastatin — Rosuvastatin
  Arms: Part 3: CC-99677, Midazolam, Digoxin, Metformin, Rosuvastatin

SUMMARY:
It is a phase 1, open-label, single-center, three-part study to assess the safety, tolerability, and pharmacokinetics of multiple doses of CC-99677 administered alone or in combination with either methotrexate and sulfasalazine; itraconazole, rifampin, midazolam, or a cocktail of digoxin, metformin, and rosuvastatin in healthy subjects

DETAILED DESCRIPTION:
This study will allow investigation of potential drug-drug interaction mediated through cytochrome P450 enzymes and drug transporter proteins. During each part, blood samples will be collected at prespecified times for pharmacokinetic assessments. Subject safety will be monitored throughout the study. There will be approximately 16 subjects enrolled into each part.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be enrolled in the study:

1. Subject is ≥ 18 and ≤ 64 years of age at the time of signing the informed consent form (ICF).

   1. Part 1 is open to male subjects ONLY
   2. Both male and female subjects may participate in Parts 2-3.
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health, as determined by the Investigator based on a physical examination at screening.
5. Female subjects of childbearing potential (FCBP) are not permitted in Part 1, but are permitted in Parts 2 and 3, and must:

   1. Have two (2) negative pregnancy tests as verified by the Investigator prior to the first dose of IP. She must agree to ongoing pregnancy testing during the course of the study, and prior to discharge from the study site. This applies even if the subject practices true abstinence2 from heterosexual contact.
   2. Agree to use, and be able to comply with, one highly effective3 non-hormonal method of contraception without interruption, during the study (including any dose interruptions), and for at least 28 days after discontinuation of IP. The female subject's chosen form of highly effective contraception must be effective by the time the female subject is enrolled into the study (eg, contraception should be initiated at least 28 days prior to enrollment) and at least 28 days after discontinuation of IP.
6. Female subjects NOT of childbearing potential are permitted in all Parts except Part 1, and must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation is required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   1. For Part 1: Agree to use a latex or other synthetic condom during sexual contact with a pregnant female or a FCBP while participating in the study, during any dose interruptions, and for at least -6 months after discontinuation of methotrexate (Methotrexate Summary of Product Characteristics [SmPC]; CTFG, 2014). In addition, any non-pregnant FCBP partner of a male subject must use a reliable contraception method, without interruption, during the study (including any dose interruptions) and for at least 6 months after discontinuation of methotrexate (Methotrexate SmPC). It is recommended that non-pregnant FCBP partners of male subjects in Part 1 use approved highly effective contraception as a reliable method. Examples of approved methods of highly effective contraception include combined hormonal contraception; progestogen only oral hormonal contraception; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomized male partner (CTFG, 2014).
   2. For Parts 2 and 3: Agree to use a latex or other synthetic condom during sexual contact with a pregnant female or a FCBP while participating in the study, during any dose interruptions, and for at least 28 days after discontinuation of IP, even if he has undergone a successful vasectomy. In addition, any non-pregnant FCBP partner of a male subject must use an approved method of effective contraception, without interruption, during the study (including any dose interruptions) and for at least 28 days after discontinuation of IP (CTFG, 2014). Examples of approved methods of effective contraception for non-pregnant FCBP partners include progestogen only oral hormonal contraception; male or female condom with or without spermicide; or cap, diaphragm, or sponge with spermicide.
8. Subject has a body mass index (BMI) ≥ 18 and ≤ 30 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. In addition, ALT, AST, and total bilirubin must be ≤ the upper limit of normal at screening and on Day -1. Platelet count, absolute neutrophil count (ANC), and absolute lymphocyte count (ALC) must be ≥ the lower limit of normal at screening and on Day -1.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has normal or clinically acceptable 12 lead ECG. In addition:

    1. If female, subject has a QTcF value ≤ 450 msec at screening.
    2. If male, subject has a QTcF value ≤ 430 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition (including but not limited to neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Female subjects are prohibited from participating in Part 1. Female subjects may participate in Parts 2-3.
5. Subject is pregnant or breastfeeding.
6. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
7. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days prior to the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer). Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
8. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration. Exceptions may apply on a case-by-case basis if considered not to interfere with the study objectives as agreed to by the Investigator and Sponsor's Medical Monitor.
9. Subject has used Cytochrome P450 (CYP) 3A inducers and/or inhibitors (including St. John's Wort) within 30 days preceding the first dose administration. The Indiana University (2016) "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP3A (http://medicine.iupui.edu/clinpharm/ddis/table.aspx). The Sponsor's Medical Monitor or designee should be queried in case of uncertainty.
10. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, or excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable. Other previous surgeries may be acceptable with concurrence of the Sponsor's Medical Monitor.
11. Subject donated blood or serum within 8 weeks before the first dose administration to a blood bank or blood donation center.
12. Subject has a history of drug abuse (as defined by the current version of the International Classification of Diseases (ICD V11.0)) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
13. Subject has a history of alcohol abuse (as defined by the NHS alcohol tracker https://www.nhs.uk/live-well/alcohol-support/calculating-alcohol-units/) within 2 years before the first dose administration, or positive alcohol screen.
14. Subject is known to have a history of hepatitis B and/or hepatitis C, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

    a. Note: Subjects who received hepatitis B vaccination and who test positive for hepatitis B surface antibody and negative for both hepatitis B surface antigen and hepatitis B core antibody remain eligible for study participation.
15. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
16. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to the first dose administration or is planning to receive immunization with a live or live attenuated vaccine for 2 months following the last dose administration.
17. Subject has a history of Gilbert's syndrome or has laboratory findings at screening that, in the opinion of the Investigator, are indicative of Gilbert's syndrome.
18. Subject has a history of incompletely treated Mycobacterium tuberculosis (TB) infection, as indicated by:

    1. Subject's medical records documenting incomplete treatment for Mycobacterium TB.
    2. Subject's self-reported history of incomplete treatment for Mycobacterium TB.
    3. Note: Subjects with a history of TB who have undergone treatment accepted by the local health authorities (documented) may be eligible for study entry.
19. Subject is part of the study site staff personnel or a family member of the study site staff.
20. Subject has previously been exposed to CC-99677 (eg in a prior clinical trial).
21. Subject has a history of photosensitivity to medications.
22. Subject has a documented allergy or history of adverse reaction to required medications in the Part for which he/she is seeking to be enrolled, specifically:

    1. Methotrexate and/or sulfasalazine (or its analogues) for Part 1
    2. Itraconazole and/or rifampin (or its analogues) for Part 2
    3. Midazolam and/or digoxin and/or metformin and/or rosuvastatin (or other HMG-CoA reductases i.e. "statins") for Part 3

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics-Cmax | Up to approximately 72 hours
  Maximum observed plasma concentration
Pharmacokinetics-AUC0-t | Up to approximately 72 hours
  Area under the plasma concentration-time curve from time zero extrapolated to the last quantifiable concentration

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of treatment
  Number of subjects with adverse events
Pharmacokinetics-Cmax | Up to approximately 72 hours
  Maximum observed plasma concentrations of metabolites
Pharmacokinetics-AUC0-t | Up to approximately 72 hours
  Ratio of area under the plasma concentration-time curve from time zero extrapolated to the last quantifiable concentration of parent and metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Kofi Mensah, MD, PhD, Study Director — Celgene
Locations (1):
- Richmond Pharmacology Limited, London, United Kingdom